CLINICAL TRIAL: NCT02310035
Title: Observational Study on the Course of Plasma Glutamine Levels During Critial Illness
Brief Title: Observational Study on the Course of Plasma Glutamine Levels During Critical Illness
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: nWMO48
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Glutamine Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood sampled for standard evaluation will be used for determination of plasma glutamine by Bioprofile Flex Glutamine Sensor at ICU admission

DETAILED DESCRIPTION:
All patients who are admitted to the ICU after elective surgery and non-elective admissions. In both groups a total of 80 patients will be included.

(In the trials we mentioned in the introduction 80, 174 and 66 patients were included. In the study performed by Oudemans-van Straaten a decent distribution between lower and higher levels of glutamine was achieved in 80 non-elective patients.) Exclusion criteria are patients younger then 18 years and patients who need total parenteral nutrition (TPN).

The patients will receive standard care during their treatment on the ICU. Blood sampled for standard evaluation will be used for determination of plasma glutamine by Bioprofile Flex Glutamine Sensor at ICU admission. Hereafter plasma glutamine will be measured daily, a plasma sample will be taken from a standard evaluation blood sample at 6.00 am during admission on the ICU.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU

Exclusion Criteria:

* younger then 18 years and patients who need total parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are admitted to the ICU after elective surgery and non-elective admissions
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
glutamine in serum | from admission up to 8 days
  glutamine level at admission and during ICU stay daily

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

REFERENCES:
- [Derived] Buter H, Bakker AJ, Kingma WP, Koopmans M, Boerma EC. Plasma glutamine levels in patients after non-elective or elective ICU admission: an observational study. BMC Anesthesiol. 2016 Mar 10;16:15. doi: 10.1186/s12871-016-0180-7. PMID 26965168